CLINICAL TRIAL: NCT06026761
Title: Validation of Myant Skiin Smart Garments for Metabolic Rate Estimation
Brief Title: Validation of Smart Garments for Metabolic Rate Estimation
Status: Completed | Type: Observational
Sponsor: Myant Medical Corp. (Industry)
Collaborators: University of Waterloo (Other)
Responsible Party: Sponsor
Other Study IDs: Myant/Waterloo/44441
Record Dates: First submitted 2023-05-23; First posted 2023-09-07 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Healthy
Keywords: wearable; metabolic; MET minute; calories; physical activity; accelerometer; heart rate
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy individuals: Metabolic study protocol
  Interventions: Device: Skiin garment and pods

INTERVENTIONS:
Device: Skiin garment and pods — Participants will be asked to wear two pieces of equipment to record physiological data:
  1. A Skiin garment that contains IMU and ECG sensors
  2. A Cosmed K5 metabolic cart that will record breathing rate data
  Participants will then be asked to perform various tasks of daily living (e.g. watching TV, sweeping the floor), general strength exercises (e.g. squats, triceps dips, lunges), and aerobic exercises (e.g. walking, running) as instructed by researchers

SUMMARY:
The goal of this observational study is to assess the use of Myant Skiin garments for the purpose of estimating metabolic rate in 20 adult (18-64 yrs) healthy participants. The main question it aims to answer is What is the accuracy of metabolic rate estimate from the Skiin algorithm utilizing Skiin data, as compared to observation and a gold-standard sensor?

Participants will be asked to perform a number of scripted tasks and their data will be assessed and compared against gold standard wearable indirect calorimetry device (COSMED K5) measurements.

.

DETAILED DESCRIPTION:
1. Following consent, the participants will first be asked to fill out a participant information questionnaire.
2. Equipment setup - SKIIN: For the SKIIN garments, participants will use the elastic research belt for the study. The belt is an fabric, elastic strap that has been washed and sanitized to be worn over the skin at the chest or waist. A private area for changing will be provided. The SKIIN sensor pod will be attached to the holster on the belt to collect inertial measurement unit (IMU) data and electrocardiography (ECG) data similar to the motion and cardiac sensors in many wrist-worn activity tracking systems (e.g., Apple Watch). The electrodes must be in contact with the skin to acquire ECG data. Data from the Skiin garments will be acquired using the custom research interface provided by the supplier. The data is acquired wirelessly and stored on the local computer (and no data is sent to the cloud).
3. Equipment setup - K5 COSMED: For the reference/criterion- standard metabolic measurement system, a wearable indirect calorimetry system will be used. This system comprises of a mask fitted over the mouth and nose connected to a portable device that analyzes breath gas composition and volume. The mask has been cleaned and sanitized prior to use with a participant. The data is acquired on the device and stored on a local computer (no data is sent to the cloud).
4. Once the equipment has been set up for the participant, an overview of the activities and exercise tasks to be conducted during the protocol will be demonstrated.
5. Exercise tasks are described in more detail in the attached document. In general, all exercises can be modified by the participant to modulate intensity

ELIGIBILITY:
Inclusion Criteria:

- Healthy male and female adult volunteers (18y - 64y old)

must answer No to the following:

* Have you had musculoskeletal and/or neurological foot, ankle, knee, or hip conditions, such as stroke, arthritis, trauma, joint surgery?
* Have you been diagnosed with a neurological disorder or cognitive impairment such as Alzheimer's disease, migraine, epilepsy, dementia, Parkinson's disease, brain tumors, multiple sclerosis?
* Have you experienced a diagnosed concussion or brain trauma in the past 6 months?
* Do you have a condition that limits your capacity for aerobic exercise (e.g., asthma, cardiac condition)?

Exclusion Criteria:

* individuals with (self-reported) lower limb conditions, neurological disorders, history of concussion/brain trauma, and/or condition limiting exercise is to mitigate additional risk for injury and/or adverse reactions associated with exercise activities.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 20 (18-64 yrs) healthy participants will be recruited as a convenience sample to validate the proposed methods. An n=20 was chosen to permit a breadth of personal characteristics regarding gait patterns and balance control behaviour.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Heart rate | Through study completion (1 hour total), average heart rate calculated every 1 minute
  Heart rate obtained via ECG from the Skiin device
Metabolic rate | Through study completion (1 hour total), average metabolic rate calculated every 1 minute
  Metabolic rate obtained via the gold standard portable metabolic cart (COSMED K5)
Acceleration /Activity counts | Through study completion (1 hour total), average activity calculated every 1 minute
  Epoch-based physical activity counts using accelerometer data obtained through Skiin device

SECONDARY OUTCOMES:
Age | During participant inclusion
  Participant age
Sex | During participant inclusion
  Participant sex (male, female, other)
Weight | During participant inclusion
  Participant weight (kg)
Height | During participant inclusion
  Participant height (cm)
Fitness Level | During participant inclusion
  Participant self-reported fitness level (sedentary, low, moderate, high, very high)

CONTACTS AND LOCATIONS:
Overall Officials: James Tung, PhD, Principal Investigator — Waterloo University
Locations (1):
- University of Waterloo - Engineering 7, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Follow data use agreement policy as outlined by Myant (de-identified data only)